CLINICAL TRIAL: NCT00881530
Title: A 78 Week Open Label Extension to Trials Assessing the Safety and Efficacy of BI 10773 as Monotherapy or in Combination With Metformin in Type 2 Diabetic Patients
Brief Title: Empagliflozin (BI 10773) in Type Two Diabetes (T2D) Patients, Open Label Extension
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1245.24; 2008-007938-21 (EudraCT Number: EudraCT)
Record Dates: First submitted 2009-04-14; First posted 2009-04-15 (Estimated); Results first posted 2014-06-16 (Estimated); Last update posted 2014-06-16 (Estimated); Status verified 2014-05

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — empagliflozin; Metformin; Sitagliptin Phosphate

ARMS (4):
- Sitagliptin (Active Comparator): 100 mg
  Interventions: Drug: Sitagliptin
- Metformin (Active Comparator): 2000 mg
  Interventions: Drug: Metformin
- BI 10773 X mg (Experimental): lower dose
  Interventions: Drug: BI 10773
- BI 10773 Y mg (Experimental): higher dose
  Interventions: Drug: BI 10773

INTERVENTIONS:
Drug: BI 10773 — BI 10773 high dose once daily
  Arms: BI 10773 Y mg
Drug: Metformin — open label comparator
  Arms: Metformin
Drug: BI 10773 — BI 10773 low dose once daily
  Arms: BI 10773 X mg
Drug: Sitagliptin — open label comparator
  Arms: Sitagliptin

SUMMARY:
The objective of the current study is to investigate the safety and efficacy of BI 10773 in 2 different doses compared to Metformin or to Sitagliptin given for 78 weeks in different modalities of treatment in patients with type 2 diabetes mellitus.

ELIGIBILITY:
Inclusion criteria:

* patients completing one of double blind phase II trials 1245.9 or 1245.10
* informed consent

Exclusion criteria:

* patients meeting withdrawal criteria of preceding trial
* significant hepatic impairment
* significant renal impairment with creatinine clearance < 50 ml/min
* contraindication to Metformin for all patients treated with Metformin
* premenopausal women that are nursing or pregnant or not practicing acceptable methods of birth control
* drug or alcohol abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 660 (Actual)
Dates: Start 2009-03; Primary Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (137):
- United States (12):
  - 1245.24.101001 Boehringer Ingelheim Investigational Site, Mission Viejo, California
  - 1245.24.101028 Boehringer Ingelheim Investigational Site, Spring Valley, California
  - 1245.24.101027 Boehringer Ingelheim Investigational Site, Walnut Creek, California
  - 1245.24.101004 Boehringer Ingelheim Investigational Site, Clearwarter, Florida
  - 1245.24.101005 Boehringer Ingelheim Investigational Site, Miami, Florida
  - 1245.24.101024 Boehringer Ingelheim Investigational Site, Saint Cloud, Florida
  - 1245.24.101014 Boehringer Ingelheim Investigational Site, Roswell, Georgia
  - 1245.24.101016 Boehringer Ingelheim Investigational Site, Staten Island, New York
  - 1245.24.101006 Boehringer Ingelheim Investigational Site, Wadsworth, Ohio
  - 1245.24.101023 Boehringer Ingelheim Investigational Site, Norristown, Pennsylvania
  - 1245.24.101015 Boehringer Ingelheim Investigational Site, Dallas, Texas
  - 1245.24.101025 Boehringer Ingelheim Investigational Site, Federal Way, Washington
- Austria (3):
  - 1245.24.431002 Boehringer Ingelheim Investigational Site, Graz
  - 1245.24.431001 Boehringer Ingelheim Investigational Site, Vienna
  - 1245.24.431003 Boehringer Ingelheim Investigational Site, Vienna
- Croatia (4):
  - 1245.24.385104 Boehringer Ingelheim Investigational Site, Karlovac
  - 1245.24.385103 Boehringer Ingelheim Investigational Site, Krapinske Toplice
  - 1245.24.385106 Boehringer Ingelheim Investigational Site, Osijek
  - 1245.24.385101 Boehringer Ingelheim Investigational Site, Zagreb
- Czechia (4):
  - 1245.24.420103 Boehringer Ingelheim Investigational Site, Brno
  - 1245.24.420105 Boehringer Ingelheim Investigational Site, Brno
  - 1245.24.420101 Boehringer Ingelheim Investigational Site, Břeclav
  - 1245.24.420102 Boehringer Ingelheim Investigational Site, Hodonín
- Estonia (5):
  - 1245.24.372101 Boehringer Ingelheim Investigational Site, Tallinn
  - 1245.24.372102 Boehringer Ingelheim Investigational Site, Tallinn
  - 1245.24.372103 Boehringer Ingelheim Investigational Site, Tallinn
  - 1245.24.372104 Boehringer Ingelheim Investigational Site, Tallinn
  - 1245.24.372105 Boehringer Ingelheim Investigational Site, Tartu
- Finland (4):
  - 1245.24.581006 Boehringer Ingelheim Investigational Site, Kerava
  - 1245.24.581003 Boehringer Ingelheim Investigational Site, Oulu
  - 1245.24.581004 Boehringer Ingelheim Investigational Site, Tampere
  - 1245.24.581001 Boehringer Ingelheim Investigational Site, Turku
- France (13):
  - 1245.24.3302A Boehringer Ingelheim Investigational Site, Bondy
  - 1245.24.3302B Boehringer Ingelheim Investigational Site, Bondy
  - 1245.24.3310A Boehringer Ingelheim Investigational Site, Caen
  - 1245.24.3310C Boehringer Ingelheim Investigational Site, Caen
  - 1245.24.3301A Boehringer Ingelheim Investigational Site, Corbeil-Essonnes
  - 1245.24.3303A Boehringer Ingelheim Investigational Site, La Rochelle
  - 1245.24.3303B Boehringer Ingelheim Investigational Site, La Rochelle
  - 1245.24.3309A Boehringer Ingelheim Investigational Site, Nanterre
  - 1245.24.3306A Boehringer Ingelheim Investigational Site, Narbonne
  - 1245.24.3304A Boehringer Ingelheim Investigational Site, Reims
  - 1245.24.3311B Boehringer Ingelheim Investigational Site, Saint-Mandé
  - 1245.24.3305A Boehringer Ingelheim Investigational Site, Valenciennes
  - 1245.24.3305B Boehringer Ingelheim Investigational Site, Valenciennes
- Germany (9):
  - 1245.24.491011 Boehringer Ingelheim Investigational Site, Aschaffenburg
  - 1245.24.491007 Boehringer Ingelheim Investigational Site, Frankfurt am Main
  - 1245.24.491004 Boehringer Ingelheim Investigational Site, Hamburg
  - 1245.24.491005 Boehringer Ingelheim Investigational Site, Hamburg
  - 1245.24.491002 Boehringer Ingelheim Investigational Site, Melsungen
  - 1245.24.491012 Boehringer Ingelheim Investigational Site, Nuremberg
  - 1245.24.491008 Boehringer Ingelheim Investigational Site, Rehlingen-Siersburg
  - 1245.24.491003 Boehringer Ingelheim Investigational Site, Saint Ingbert/Oberwürzbach
  - 1245.24.491010 Boehringer Ingelheim Investigational Site, Sulzbach-Rosenberg
- Hungary (5):
  - 1245.24.361001 Boehringer Ingelheim Investigational Site, Budapest
  - 1245.24.361003 Boehringer Ingelheim Investigational Site, Budapest
  - 1245.24.361004 Boehringer Ingelheim Investigational Site, Budapest
  - 1245.24.361005 Boehringer Ingelheim Investigational Site, Győr
  - 1245.24.361002 Boehringer Ingelheim Investigational Site, Szombathely
- Italy (3):
  - 1245.24.391006 Boehringer Ingelheim Investigational Site, Genova
  - 1245.24.391003 Boehringer Ingelheim Investigational Site, Pisa
  - 1245.24.391005 Boehringer Ingelheim Investigational Site, Treviso
- Latvia (7):
  - 1245.24.371101 Boehringer Ingelheim Investigational Site, Daugavpils
  - 1245.24.371105 Boehringer Ingelheim Investigational Site, Kuldīga
  - 1245.24.371106 Boehringer Ingelheim Investigational Site, Ogre
  - 1245.24.371103 Boehringer Ingelheim Investigational Site, Riga
  - 1245.24.371107 Boehringer Ingelheim Investigational Site, Riga
  - 1245.24.371102 Boehringer Ingelheim Investigational Site, Talsi
  - 1245.24.371104 Boehringer Ingelheim Investigational Site, Valmiera
- Lithuania (2):
  - 1245.24.370102 Boehringer Ingelheim Investigational Site, Klaipėda
  - 1245.24.370101 Boehringer Ingelheim Investigational Site, Vilnius
- Norway (4):
  - 1245.24.471004 Boehringer Ingelheim Investigational Site, Ålesund
  - 1245.24.471003 Boehringer Ingelheim Investigational Site, Hamar
  - 1245.24.471005 Boehringer Ingelheim Investigational Site, Oslo
  - 1245.24.471001 Boehringer Ingelheim Investigational Site, Stavanger
- Romania (8):
  - 1245.24.401005 Boehringer Ingelheim Investigational Site, Alba Iulia
  - 1245.24.401006 Boehringer Ingelheim Investigational Site, Baia Mare Maramures
  - 1245.24.401002 Boehringer Ingelheim Investigational Site, Brasov
  - 1245.24.401001 Boehringer Ingelheim Investigational Site, Bucharest
  - 1245.24.401008 Boehringer Ingelheim Investigational Site, Bucharest
  - 1245.24.401003 Boehringer Ingelheim Investigational Site, Galati
  - 1245.24.401007 Boehringer Ingelheim Investigational Site, Satu Mare
  - 1245.24.401004 Boehringer Ingelheim Investigational Site, Târgu Mureş
- Russia (12):
  - 1245.24.701002 Boehringer Ingelheim Investigational Site, Kazan'
  - 1245.24.701008 Boehringer Ingelheim Investigational Site, Moscow
  - 1245.24.701009 Boehringer Ingelheim Investigational Site, Moscow
  - 1245.24.701010 Boehringer Ingelheim Investigational Site, Moscow
  - 1245.24.701004 Boehringer Ingelheim Investigational Site, Petrozavodsk
  - 1245.24.701012 Boehringer Ingelheim Investigational Site, Saint Petersburg
  - 1245.24.701013 Boehringer Ingelheim Investigational Site, Saint Petersburg
  - 1245.24.701014 Boehringer Ingelheim Investigational Site, Saratov
  - 1245.24.701005 Boehringer Ingelheim Investigational Site, Smolensk
  - 1245.24.701006 Boehringer Ingelheim Investigational Site, Yaroslavl
  - 1245.24.701007 Boehringer Ingelheim Investigational Site, Yaroslavl
  - 1245.24.701001 Boehringer Ingelheim Investigational Site, Yekaterinburg
- Slovakia (8):
  - 1245.24.421102 Boehringer Ingelheim Investigational Site, Bratislava
  - 1245.24.421107 Boehringer Ingelheim Investigational Site, Bratislava
  - 1245.24.421103 Boehringer Ingelheim Investigational Site, Lučenec
  - 1245.24.421105 Boehringer Ingelheim Investigational Site, Nitra
  - 1245.24.421106 Boehringer Ingelheim Investigational Site, Nitra
  - 1245.24.421104 Boehringer Ingelheim Investigational Site, Nové Mesto nad Váhom
  - 1245.24.421108 Boehringer Ingelheim Investigational Site, Prešov
  - 1245.24.421101 Boehringer Ingelheim Investigational Site, Prievidza
- South Korea (8):
  - 1245.24.821006 Boehringer Ingelheim Investigational Site, Goyang
  - 1245.24.821008 Boehringer Ingelheim Investigational Site, Goyang
  - 1245.24.821007 Boehringer Ingelheim Investigational Site, Incheon
  - 1245.24.821002 Boehringer Ingelheim Investigational Site, Pucheon
  - 1245.24.821001 Boehringer Ingelheim Investigational Site, Seoul
  - 1245.24.821004 Boehringer Ingelheim Investigational Site, Seoul
  - 1245.24.821009 Boehringer Ingelheim Investigational Site, Suwon
  - 1245.24.821003 Boehringer Ingelheim Investigational Site, Uijeongbu-si
- Spain (7):
  - 1245.24.341002 Boehringer Ingelheim Investigational Site, Barcelona
  - 1245.24.341001 Boehringer Ingelheim Investigational Site, Girona
  - 1245.24.341010 Boehringer Ingelheim Investigational Site, L'Hospitalet de Llobregat (Barcelona)
  - 1245.24.341004 Boehringer Ingelheim Investigational Site, Málaga
  - 1245.24.341005 Boehringer Ingelheim Investigational Site, Palma Mallorca
  - 1245.24.341006 Boehringer Ingelheim Investigational Site, Palma Mallorca
  - 1245.24.341008 Boehringer Ingelheim Investigational Site, Santander
- Sweden (3):
  - 1245.24.461004 Boehringer Ingelheim Investigational Site, Härnösand
  - 1245.24.461005 Boehringer Ingelheim Investigational Site, Lund
  - 1245.24.461001 Boehringer Ingelheim Investigational Site, Stockholm
- Taiwan (7):
  - 1245.24.886105 Boehringer Ingelheim Investigational Site, Changhua
  - 1245.24.886107 Boehringer Ingelheim Investigational Site, Kaohsiung City
  - 1245.24.886104 Boehringer Ingelheim Investigational Site, Taichun
  - 1245.24.886106 Boehringer Ingelheim Investigational Site, Tainan
  - 1245.24.886101 Boehringer Ingelheim Investigational Site, Taipei
  - 1245.24.886103 Boehringer Ingelheim Investigational Site, Taipei
  - 1245.24.886102 Boehringer Ingelheim Investigational Site, Taoyuan District
- Ukraine (9):
  - 1245.24.381007 Boehringer Ingelheim Investigational Site, Dnipro
  - 1245.24.381003 Boehringer Ingelheim Investigational Site, Kharkiv
  - 1245.24.381009 Boehringer Ingelheim Investigational Site, Kharkiv
  - 1245.24.381010 Boehringer Ingelheim Investigational Site, Kharkiv
  - 1245.24.381008 Boehringer Ingelheim Investigational Site, Kiev
  - 1245.24.381002 Boehringer Ingelheim Investigational Site, Odesa
  - 1245.24.381006 Boehringer Ingelheim Investigational Site, Vinnitsa
  - 1245.24.381001 Boehringer Ingelheim Investigational Site, Vinnytsia
  - 1245.24.381005 Boehringer Ingelheim Investigational Site, Vinnytsia

REFERENCES:
- [Derived] Ferrannini E, Berk A, Hantel S, Pinnetti S, Hach T, Woerle HJ, Broedl UC. Long-term safety and efficacy of empagliflozin, sitagliptin, and metformin: an active-controlled, parallel-group, randomized, 78-week open-label extension study in patients with type 2 diabetes. Diabetes Care. 2013 Dec;36(12):4015-21. doi: 10.2337/dc13-0663. Epub 2013 Nov 1. PMID 24186878

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was an open label extension trial of the blinded 12-week dose-finding studies NCT00789035 and NCT00749190.
Pre-assignment Details: Patients from the preceding empagliflozin 10 and 25 mg groups continued to take the same doses. Patients on placebo and other empagliflozin doses were re-randomised to one of the empagliflozin treatments. Patients on metformin monotherapy or sitagliptin added-on to metformin in the preceding trials continued their open label treatments.
Groups:
- Empagliflozin 10 mg: Patients receive 10 mg Empagliflozin in tablets once daily.
- Empagliflozin 25 mg: Patients receive 25 mg Empagliflozin in tablets once daily.
- Metformin: Patients receive between 1000 and 2000 mg Metformin daily as monotherapy. Patients on metformin as active comparator (from trial NCT00789035) were to take their medication according to the instruction of their investigator, continuing the maximum tolerated dose determined in the preceding trial.
- Empagliflozin 10 mg + Metformin: Patients receive 10 mg Empagliflozin in tablets once daily added to metformin background. Patients on metformin background (from trial NCT00749190) continued with their standard metformin therapy throughout the entire study.
- Empagliflozin 25 mg + Metformin: Patients receive 25 mg Empagliflozin in tablets once daily added to metformin background. Patients on metformin background (from trial NCT00749190) continued with their standard metformin therapy throughout the entire study.
- Sitaglipin + Metformin: Patients receive 100 mg Sitagliptin once daily in tablets added to metformin background. Patients on metformin background (from trial NCT00749190) continued with their standard metformin therapy throughout the entire study.
Period: Overall Study
Arm/Group | Empagliflozin 10 mg | Empagliflozin 25 mg | Metformin | Empagliflozin 10 mg + Metformin | Empagliflozin 25 mg + Metformin | Sitaglipin + Metformin
Started | 106 | 109 | 56 | 166 | 166 | 56
Completed | 92 | 104 | 51 | 157 | 152 | 51
Not Completed | 14 | 5 | 5 | 9 | 14 | 5
Not completed — Adverse Event | 5 | 1 | 1 | 4 | 10 | 2
Not completed — Lack of Efficacy | 1 | 0 | 0 | 0 | 1 | 1
Not completed — Not compliant with the protocol | 0 | 0 | 0 | 0 | 2 | 0
Not completed — Lost to Follow-up | 0 | 1 | 1 | 3 | 1 | 0
Not completed — Refused to continue medication | 7 | 2 | 1 | 2 | 0 | 0
Not completed — Other reason not defined above | 1 | 1 | 2 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Population: Treated set including all patients treated with at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Empagliflozin 10 mg | Empagliflozin 25 mg | Metformin | Empagliflozin 10 mg + Metformin | Empagliflozin 25 mg + Metformin | Sitaglipin + Metformin | Total
Number analyzed (Participants) | 106 | 109 | 56 | 166 | 166 | 56 | 659
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.3 (8.5) | 58.5 (10.0) | 56.8 (8.9) | 58.4 (8.3) | 59.9 (7.8) | 58.3 (10.5) | 58.6 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57 | 52 | 28 | 83 | 78 | 27 | 325
  Male | 49 | 57 | 28 | 83 | 88 | 29 | 334

OUTCOME MEASURES:

1. Primary Outcome: Hypoglycaemic Events
Description: Investigator defined Hypoglycaemic events. For documentation of hypoglycemic events, the following criteria were taken into consideration:
  * Asymptomatic hypoglycemia: the event was not accompanied by typical symptoms of hypoglycemia but with a measured plasma glucose of ≤70 mg/dL (≤3.9 mmol/L)
  * Documented symptomatic hypoglycemia with glucose of ≥54 mg/dL and ≤70 mg/dL (≥3.0 mmol/L and ≤3.9 mmol/L)
  * Documented symptomatic hypoglycemia with glucose of <54 mg/dL (<3.0 mmol/L): the event was accompanied by typical symptoms of hypoglycemia but in no need for external assistance
  * Severe hypoglycemic episode: the event required the assistance of another person to actively administer carbohydrate, glucagon, or other resuscitative actions
Time Frame: 78 weeks plus 1 week of follow-up
Population: Treated set
Measure: Number; unit: percentage of participants
Arm/Group | Empagliflozin 10 mg | Empagliflozin 25 mg | Metformin | Empagliflozin 10 mg + Metformin | Empagliflozin 25 mg + Metformin | Sitaglipin + Metformin
Number analyzed (Participants) | 106 | 109 | 56 | 166 | 166 | 56
percentage of participants | 0.9 | 1.8 | 7.1 | 2.4 | 3.6 | 5.4

2. Primary Outcome: Change From Baseline to Week 78 in Lipid Parameters
Description: Change from baseline to week 78 in lipid parameters (Total cholesterol, High-density lipoprotein (HDL), Low-density lipoprotein (LDL) and Triglyceride)
Time Frame: Weeks 1 and 78
Population: Treated set
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Empagliflozin 10 mg | Empagliflozin 25 mg | Metformin | Empagliflozin 10 mg + Metformin | Empagliflozin 25 mg + Metformin | Sitaglipin + Metformin
Number analyzed (Participants) | 105 | 109 | 56 | 164 | 162 | 56
mmol/L
  Total Cholesterol | -0.13 (1.17) | 0.09 (0.88) | -0.24 (0.77) | 0.19 (0.81) | 0.13 (0.75) | -0.05 (0.91)
  HDL | 0.08 (0.11) | 0.07 (0.10) | 0.06 (0.10) | 0.06 (0.09) | 0.07 (0.10) | 0.03 (0.08)
  LDL (N=102, 108, 52, 161, 159, 55) | -0.02 (0.83) | 0.05 (0.83) | -0.13 (0.74) | 0.13 (0.71) | 0.07 (0.69) | 0.00 (0.79)
  Triglyceride | -0.5 (2.3) | -0.0 (0.6) | -0.5 (1.2) | 0.1 (0.9) | -0.1 (0.8) | -0.2 (0.9)

3. Secondary Outcome: Change From Baseline in HbA1c Over Time
Description: Baseline source: before first intake of active treatment (preceding trial or Open label extension)
Time Frame: Weeks 1, 6, 18, 30, 42, 54, 66 and 78
Population: Treated set
Measure: Mean (Standard Deviation); unit: percentage of HbA1c
Arm/Group | Empagliflozin 10 mg | Empagliflozin 25 mg | Metformin | Empagliflozin 10 mg + Metformin | Empagliflozin 25 mg + Metformin | Sitaglipin + Metformin
Number analyzed (Participants) | 106 | 109 | 56 | 166 | 166 | 56
percentage of HbA1c
  Week 6 (N=104, 108, 55, 162, 163, 54) | -0.40 (0.77) | -0.57 (0.81) | -1.03 (0.76) | -0.36 (0.67) | -0.55 (0.60) | -0.75 (0.80)
  Week 18 (N=93, 105, 53, 149, 157, 48) | -0.58 (0.75) | -0.72 (0.88) | -0.92 (0.91) | -0.51 (0.68) | -0.70 (0.68) | -0.79 (0.84)
  Week 30 (N=93, 99, 50, 140, 151, 45) | -0.47 (0.85) | -0.61 (0.90) | -0.95 (0.82) | -0.58 (0.69) | -0.76 (0.70) | -0.68 (0.82)
  Week 42 (N=85, 93, 46, 132, 140, 44) | -0.59 (0.87) | -0.74 (0.98) | -1.10 (0.80) | -0.65 (0.72) | -0.79 (0.76) | -0.51 (1.03)
  Week 54 (N=78, 85, 44, 128, 136, 41) | -0.66 (0.83) | -0.71 (0.87) | -1.13 (0.89) | -0.62 (0.76) | -0.75 (0.73) | -0.79 (0.79)
  Week 66 (N=80, 87, 43, 120, 127, 39) | -0.55 (0.80) | -0.71 (1.01) | -1.04 (0.79) | -0.59 (0.79) | -0.73 (0.77) | -0.78 (0.90)
  Week 78 (N=72, 84, 42, 115, 121, 38) | -0.50 (0.77) | -0.55 (0.90) | -0.80 (0.88) | -0.56 (0.80) | -0.71 (0.81) | -0.66 (0.99)

4. Secondary Outcome: Occurence of a Treat-to-target Response (HbA1c < 7.0%)
Description: Occurence of a treat-to-target response, defined as HbA1c < 7.0% over time
Time Frame: Weeks 1, 6, 18, 30, 42, 54, 66 and 78
Population: Treated set
Measure: Number; unit: percentage of participants
Arm/Group | Empagliflozin 10 mg | Empagliflozin 25 mg | Metformin | Empagliflozin 10 mg + Metformin | Empagliflozin 25 mg + Metformin | Sitaglipin + Metformin
Number analyzed (Participants) | 106 | 109 | 56 | 166 | 166 | 56
percentage of participants
  Week 6 (N=104, 108, 55, 162, 163, 54) | 26.9 | 25.0 | 45.5 | 24.1 | 25.2 | 35.2
  Week 18 (N=93, 105, 53, 149, 157, 48) | 33.3 | 33.3 | 45.3 | 31.5 | 37.6 | 35.4
  Week 30 (N=93, 99, 50, 140, 151, 45) | 34.4 | 29.3 | 42.0 | 28.6 | 45.7 | 28.9
  Week 42 (N=85, 93, 46, 132, 140, 44) | 41.2 | 40.9 | 52.2 | 39.4 | 47.1 | 25.0
  Week 54 (N=78, 85, 44, 128, 136, 41) | 43.6 | 32.9 | 56.8 | 35.9 | 47.8 | 29.3
  Week 66 (N=80, 87, 43, 120, 127, 39) | 31.3 | 39.1 | 44.2 | 35.8 | 48.0 | 38.5
  Week 78 (N=72, 84, 42, 115, 121, 38) | 31.9 | 32.1 | 31.0 | 27.0 | 44.6 | 36.8

5. Secondary Outcome: Occurrence of a Treat-to-target Response (HbA1c < 6.5%)
Description: Occurrence of a Treat-to-target Response, defined as HbA1c < 6.5% over time
Time Frame: Weeks 1, 6, 18, 30, 42, 54, 66 and 78
Population: Treated set
Measure: Number; unit: percentage of participants
Arm/Group | Empagliflozin 10 mg | Empagliflozin 25 mg | Metformin | Empagliflozin 10 mg + Metformin | Empagliflozin 25 mg + Metformin | Sitaglipin + Metformin
Number analyzed (Participants) | 106 | 109 | 56 | 166 | 166 | 56
percentage of participants
  Week 6 (N=104, 108, 55, 162, 163, 54) | 3.8 | 11.1 | 16.4 | 6.2 | 6.7 | 11.1
  Week 18 (N=93, 105, 53, 149, 157, 48) | 11.8 | 12.4 | 13.2 | 4.7 | 5.1 | 12.5
  Week 30 (N=93, 99, 50, 140, 151, 45) | 8.6 | 10.1 | 14.0 | 8.6 | 10.6 | 4.4
  Week 42 (N=85, 93, 46, 132, 140, 44) | 11.8 | 10.8 | 21.7 | 10.6 | 21.4 | 9.1
  Week 54 (N=78, 85, 44, 128, 136, 41) | 11.5 | 5.9 | 18.2 | 10.9 | 15.4 | 9.8
  Week 66 (N=80, 87, 43, 120, 127, 39) | 10.0 | 11.5 | 14.0 | 8.3 | 12.6 | 15.4
  Week 78 (N=72, 84, 42, 115, 121, 38) | 6.9 | 8.3 | 9.5 | 10.4 | 13.2 | 18.4

6. Secondary Outcome: Occurrence of a Relative Efficacy Response
Description: Occurrence of a Relative Efficacy Response (HbA1c Lowered by at least >=0.5% over time)
Time Frame: Weeks 1, 6, 18, 30, 42, 54, 66 and 78
Population: Treated set
Measure: Number; unit: percentage of participants
Arm/Group | Empagliflozin 10 mg | Empagliflozin 25 mg | Metformin | Empagliflozin 10 mg + Metformin | Empagliflozin 25 mg + Metformin | Sitaglipin + Metformin
Number analyzed (Participants) | 106 | 109 | 56 | 166 | 166 | 56
percentage of participants
  Week 6 (N=104, 108, 55, 162, 163, 54) | 42.3 | 50.9 | 80.0 | 41.4 | 56.4 | 63.0
  Week 18 (N=93, 105, 53, 149, 157, 48) | 51.6 | 61.9 | 77.4 | 53.7 | 61.8 | 66.7
  Week 30 (N=93, 99, 50, 140, 151, 45) | 50.5 | 55.6 | 78.0 | 55.0 | 63.6 | 68.9
  Week 42 (N=85, 93, 46, 132, 140, 44) | 58.8 | 60.2 | 82.6 | 62.1 | 66.4 | 54.5
  Week 54 (N=78, 85, 44, 128, 136, 41) | 62.8 | 58.8 | 81.8 | 59.4 | 65.4 | 58.5
  Week 66 (N=80, 87, 43, 120, 127, 39) | 53.8 | 56.3 | 76.7 | 55.0 | 64.6 | 66.7
  Week 78 (N=72, 84, 42, 115, 121, 38) | 50.0 | 50.0 | 66.7 | 56.5 | 64.5 | 60.5

7. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG) Over Time
Description: Baseline source: before first intake of active treatment (preceding trial or Open label extension)
Time Frame: Weeks 1, 6, 18, 30, 42, 54, 66 and 78
Population: Treated set
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Empagliflozin 10 mg | Empagliflozin 25 mg | Metformin | Empagliflozin 10 mg + Metformin | Empagliflozin 25 mg + Metformin | Sitaglipin + Metformin
Number analyzed (Participants) | 106 | 109 | 56 | 166 | 166 | 56
mg/dL
  Week 6 (N=102, 108, 55, 156, 160, 53) | -30.6 (42.5) | -35.8 (39.6) | -29.9 (40.0) | -25.7 (35.2) | -36.7 (36.3) | -32.6 (42.4)
  Week 18 (N=94, 103, 51, 144, 153, 45) | -35.5 (37.9) | -33.7 (42.0) | -30.4 (40.3) | -30.6 (31.6) | -37.6 (35.8) | -16.7 (44.0)
  Week 30 (N=92, 101, 51, 133, 147, 43) | -32.3 (41.4) | -35.0 (39.6) | -28.5 (28.9) | -29.9 (34.9) | -37.9 (38.6) | -25.6 (38.6)
  Week 42 (N=85, 93, 46, 126, 140, 42) | -35.8 (39.1) | -31.3 (41.4) | -31.0 (35.6) | -30.8 (36.4) | -36.8 (34.1) | -18.5 (43.1)
  Week 54 (N=80, 88, 44, 124, 134, 39) | -32.1 (37.2) | -31.0 (37.8) | -31.8 (35.9) | -28.2 (33.7) | -36.8 (32.5) | -29.4 (35.4)
  Week 66 (N=80, 86, 43, 116, 125, 38) | -28.0 (41.4) | -28.6 (42.6) | -26.4 (35.7) | -21.7 (36.2) | -29.6 (36.4) | -32.5 (46.9)
  Week 78 (N=72, 84, 43, 112, 121, 36) | -27.9 (33.1) | -25.4 (40.9) | -22.9 (39.7) | -24.7 (41.5) | -31.9 (36.5) | -25.7 (48.9)

8. Primary Outcome: Clinical Relevant Abnormalities for Physical Examination, Vital Signs, ECG and Laboratory Measurements
Description: Clinical Relevant Abnormalities for Physical Examination, Vital Signs, ECG and Laboratory Measurements. New abnormal findings or worsening of baseline conditions were reported as treatment related Adverse Events.
Time Frame: 78 weeks plus 1 week of follow-up
Population: Treated set
Measure: Number; unit: percentage of participants
Arm/Group | Empagliflozin 10 mg | Empagliflozin 25 mg | Metformin | Empagliflozin 10 mg + Metformin | Empagliflozin 25 mg + Metformin | Sitaglipin + Metformin
Number analyzed (Participants) | 106 | 109 | 56 | 166 | 166 | 56
percentage of participants
  Alanine aminotransferase increased | 0.9 | 0.9 | 3.6 | 0.6 | 0.6 | 1.8
  Aspartate aminotransferase increased | 1.9 | 0.0 | 1.8 | 0.0 | 0.6 | 0.0
  Gamma-glutamyltransferase increased | 0.9 | 0.0 | 1.8 | 0.0 | 1.2 | 0.0
  Blood alkaline phosphatase increased | 0.9 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Blood creatine phosphokinase increased | 0.9 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Granulocyte count decreased | 0.9 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Hepatic enzyme increased | 0.0 | 0.9 | 0.0 | 0.6 | 0.0 | 0.0
  Blood creatinine increased | 0.9 | 0.9 | 0.0 | 0.0 | 0.6 | 0.0
  Creatinine renal clearance decreased | 0.0 | 0.0 | 0.0 | 0.6 | 0.0 | 0.0
  Weight decreased | 0.0 | 0.9 | 0.0 | 0.0 | 0.6 | 0.0
  Sick sinus syndrome | 0.9 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Tachycardia | 0.9 | 1.8 | 0.0 | 0.6 | 0.6 | 0.0

ADVERSE EVENTS:
Time Frame: From drug administration until 7 days after the last intake of study drug, up to 582 days
Arm/Group | Empagliflozin 10 mg | Empagliflozin 25 mg | Metformin | Empagliflozin 10 mg + Metformin | Empagliflozin 25 mg + Metformin | Sitaglipin + Metformin
Serious Adverse Events (participants affected / at risk) | 10/106 | 7/109 | 3/56 | 10/166 | 13/166 | 9/56
Other Adverse Events (participants affected / at risk) | 34/106 | 46/109 | 27/56 | 74/166 | 79/166 | 26/56
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Empagliflozin 10 mg (N=106) | Empagliflozin 25 mg (N=109) | Metformin (N=56) | Empagliflozin 10 mg + Metformin (N=166) | Empagliflozin 25 mg + Metformin (N=166) | Sitaglipin + Metformin (N=56)
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Anal abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Post procedural infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0
Cervix carcinoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1
Refractory cytopenia with multilineage dysplasia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0
Goitre (Endocrine disorders) | 0 | 0 | 0 | 0 | 1 | 0
Thyroid cyst (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 2
Cerebral infarction (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 2
Aphasia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hemiplegia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Ischaemic stroke (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 0 | 0 | 2 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Carotid artery stenosis (Nervous system disorders) | 0 | 0 | 0 | 1 | 1 | 0
Visual acuity reduced (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Angina unstable (Cardiac disorders) | 0 | 0 | 0 | 1 | 1 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0 | 1 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0
Coronary artery disease (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Myocardial ischaemia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Colonic polyp (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Abdominal hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Anal fistula (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Gingival cyst (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Lumbar hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 2
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 0 | 1 | 0 | 1
Bile duct obstruction (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 2 | 1 | 0 | 0 | 0 | 0
Death (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Traumatic fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 1 | 0
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Ligament rupture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Post procedural haematuria (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Vascular graft occlusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Burns second degree (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0
Meniscus lesion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0
Hysterectomy (Surgical and medical procedures) | 0 | 0 | 0 | 1 | 0 | 0
Abortion induced (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Empagliflozin 10 mg (N=106) | Empagliflozin 25 mg (N=109) | Metformin (N=56) | Empagliflozin 10 mg + Metformin (N=166) | Empagliflozin 25 mg + Metformin (N=166) | Sitaglipin + Metformin (N=56)
Nasopharyngitis (Infections and infestations) | 10 | 8 | 9 | 12 | 15 | 5
Urinary tract infection (Infections and infestations) | 3 | 4 | 1 | 12 | 18 | 5
Bronchitis (Infections and infestations) | 2 | 3 | 2 | 2 | 8 | 6
Upper respiratory tract infection (Infections and infestations) | 5 | 8 | 1 | 3 | 2 | 1
Viral infection (Infections and infestations) | 0 | 7 | 1 | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 12 | 16 | 8 | 36 | 25 | 9
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 2 | 4 | 4 | 6 | 3
Headache (Nervous system disorders) | 1 | 7 | 4 | 6 | 7 | 0
Hypertension (Vascular disorders) | 4 | 3 | 4 | 5 | 2 | 4
Nausea (Gastrointestinal disorders) | 2 | 2 | 3 | 6 | 6 | 4
Diarrhoea (Gastrointestinal disorders) | 2 | 3 | 3 | 3 | 4 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 3 | 0 | 1 | 0 | 3
Chest pain (General disorders) | 2 | 0 | 3 | 2 | 0 | 1
Fatigue (General disorders) | 0 | 1 | 1 | 1 | 1 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.